CLINICAL TRIAL: NCT00078000
Title: A Phase 2 Study Of The Efficacy And Safety Of SU011248 In Patients With Metastatic Breast Cancer
Brief Title: A Study of SU11248 In Patients With Metastatic Breast Cancer Who Have Failed Selected Other Therapies.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181002; NCT00095615 (obsolete NCT alias)
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib

INTERVENTIONS:
Drug: SU011248

SUMMARY:
Assessment of safety and efficacy of SU11248 in patients with metastatic breast cancer who have failed selected other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Anthracycline and taxane-refractory or intolerant metastatic breast cancer
* Female

Exclusion Criteria:

* Prior treatment with 3 or greater regimens of chemotherapy in the advanced/metastatic disease setting beyond those containing anthracyclines/taxanes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Anti-tumor efficacy

SECONDARY OUTCOMES:
Tumor control survival safety pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts

REFERENCES:
- [Derived] Keyvanjah K, DePrimo SE, Harmon CS, Huang X, Kern KA, Carley W. Soluble KIT correlates with clinical outcome in patients with metastatic breast cancer treated with sunitinib. J Transl Med. 2012 Aug 16;10:165. doi: 10.1186/1479-5876-10-165. PMID 22897944
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181002&StudyName=Assessment+Of+Safety+And+Efficacy+Of+SU11248+In+Patients+With+Metastatic+Breast+Cancer+Who+Have+Failed+Selected+Other+Therapies%2E++